CLINICAL TRIAL: NCT01079143
Title: Prospective, Multicenter, Randomized Open Study to Evaluate the Progression of Renal Graft Fibrosis According to the Epithelial-mesenchymal Transition (EMT) in de Novo Renal Transplant Recipients Treated Either by a CNI Free Immunosuppressive Regimen With Everolimus and Enteric-coated Mycophenolate Sodium or a CNI Based Regimen With Cyclosporine and Enteric-coated Mycophenolate Sodium
Brief Title: Progression of Renal Interstitial Fibrosis / Tubular Atrophy (IF/TA) According to Epithelial-mesenchymal Transition (EMT) and Immunosuppressive Regimen (Everolimus Based Versus CNI Based) in de Novo Renal Transplant Recipients
Acronym: CERTITEM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001AFR10; 2009-011473-33 (EudraCT Number)
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Results first posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-01

CONDITIONS: Renal Interstitial Fibrosis
Keywords: De Novo renal transplantation
MeSH Terms: interventions — Everolimus; Cyclosporine; Mycophenolic Acid; Basiliximab; Adrenal Cortex Hormones

ARMS (4):
- Certican EMT+ (Experimental): Patients randomized to the Certican® treatment group started this treatment after randomization (which took place 3 to 4 months post-transplantation), preferably in the evening, otherwise the following morning. Patients in the Neoral® treatment group did not receive Certican®.
  Interventions: Drug: Certican®; Drug: Myfortic; Drug: Simulect®; Drug: Corticosteroids
- Certican EMT- (Experimental): Patients randomized to the Certican® treatment group started this treatment after randomization (which took place 3 to 4 months post-transplantation), preferably in the evening, otherwise the following morning. Patients in the Neoral® treatment group did not receive Certican®.
  Interventions: Drug: Certican®; Drug: Myfortic; Drug: Simulect®; Drug: Corticosteroids
- Neoral EMT+ (Active Comparator): Between transplantation and randomization, all patients have received Neoral®. Treatment had to be initiated within 24 hours post-transplantation in combination with Myfortic®.
  Interventions: Drug: Neoral; Drug: Myfortic; Drug: Simulect®; Drug: Corticosteroids
- Neoral EMT- (Active Comparator): Between transplantation and randomization, all patients have received Neoral®. Treatment had to be initiated within 24 hours post-transplantation in combination with Myfortic®.
  Interventions: Drug: Neoral; Drug: Myfortic; Drug: Simulect®; Drug: Corticosteroids

INTERVENTIONS:
Drug: Certican® — Certican® was supplied to the participating centers by Novartis for the whole duration of the study in the form of tablets containing 0.75, 0.5 and 0.25 mg and packaged in blister packs.
  Other Names: Everolimus; RAD001
  Arms: Certican EMT+; Certican EMT-
Drug: Neoral — Neoral® was also supplied to participating centers for the entire duration of the study in the form of soft capsules of 10 mg, 25 mg, 50 mg and 100 mg, and packaged in blister packs.
  Other Names: Cyclosporine
  Arms: Neoral EMT+; Neoral EMT-
Drug: Myfortic — Myfortic ® was supplied to the participating centers for the duration of the study in the form of 180 and 360 mg gastro-resistant, film-coated tablets. Myfortic® treatment was provided to patients preoperatively or within 24 hours post-transplantation according to the practices of the center. The starting dose was generally 1,440 mg/day, in 2 daily oral fractions, administered at 12 hour intervals up to randomization. Depending on the practices of the center and for the first 6 weeks post-transplantation, a maximum daily dose of 2160 mg of Myfortic® could be administered. In the Neoral® group, the daily dose of 1440 mg was maintained throughout the study.
  In the Certican® group, the dose was halved (i.e. 720 mg/day) on introducing Certican® and maintained at 720 mg/day until the end of the study.
  An increase in the daily dose of Myfortic® (in the Certican® group) was not authorized unless this was a temporary increase that did not exceed a period of 14 consecutive days.
Drug: Simulect® — The administration of Simulect® was part of the standard immunosuppressant therapy. This induction therapy was provided to patients in the form of commercial ampoules each containing 20 mg. Simulect® was administered to each patient at the dose of 20 mg on D0 and D4 post-transplantation.
  Other Names: basiliximab
Drug: Corticosteroids — An intravenous steroid treatment could be administered peri or intraoperatively according to local practice at each center. Oral steroid treatment was quickly introduced (in the week following transplantation) at a daily dose of 20 mg and was then reduced and continued throughout the study at a minimum dose of 5 mg/day.

SUMMARY:
Recently, early biomarkers of renal interstitial fibrosis have been identified, amongst them de novo expression of vimentin by tubular epithelial cells, which is an intermediate filament, and the translocation of beta-catenin into their cytoplasm. These markers, when present, suggest that the epithelial cell undergoes a phenomenon well known as "epithelial to mesenchymal transition" (EMT) and could behaves like a myo-fibroblast. EMT is highly instrumental in several models of tissue fibrosis, including in the kidney. Actually, it has not only been demonstrated that these markers are detectable in the renal graft at an early time point post-transplant (i.e. as soon as three months), but also that the intensity of their expression correlates with the progression of interstitial fibrosis of the graft between 3 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a primary or secondary deceased or living (related or not) donor kidney transplant and who requires basiliximab induction therapy.
* Cold ischemia time < 30 hours.
* Women of child-bearing age, even those with a history of infertility, must have had a negative pregnancy test during the 7 days before screening or at the time of screening, and must use a recognized and reliable method of contraception throughout the study and for 2 months after discontinuing the study treatment.
* Patients who want and are able to take part in the entire study, and have given their written consent.
* Patients who are registered with a French national health insurance scheme or are covered by such a scheme.

Exclusion Criteria:

* Recipient of multi-organ transplantation, including dual kidneys, or who have previously received non renal transplant organ.
* Patients receiving a graft from a non-heart-beating donor.
* Anti-HLA antibody levels ≥ 20% in the last 3 months before the inclusion.
* ABO incompatible graft or with positive cross match T.
* Severe hyperlipidemia: total cholesterol ≥ 9.1 mmol/L (≥ 350 mg/dL) and/or triglycerides ≥ 8.5 mmol/L (≥ 750 mg/dL) despite appropriate lipid-lowering therapy.
* Known hypersensitivity or contraindications to mycophenolic acid, cyclosporine or lactose.
* Known hypersensitivity or contraindications to macrolides or drugs of the mTOR inhibitor class.
* HIV seropositive, or active chronic hepatitis B (HBs Ab) or C. Results obtained during the 6 months before the inclusion are accepted. Recipients from donors with hepatitis B or C will be excluded.
* Patients with thrombocytopenia (≤ 75000/mm3), absolute neutrophil count (≤ 1500/mm3), leukocytopenia (≤ 2500/mm3) and/or hemoglobin < 8g/dL at the inclusion visit.
* ASAT, ALAT or total bilirubin ≥ 3 UNL.
* Uncontrolled severe infection, severe allergy requiring an acute or chronic treatment.
* Patients with a malignant disease or previous malignancy in the past 5 years, with the exception of excised basal cell or squamous cell carcinoma and in situ cervical cancer treated.
* Medical or surgical condition, with the exception of the transplantation, which in the investigator's opinion could exclude the patient.
* Women who are pregnant, breastfeeding or of reproductive age and refuse or are unable to use a recognized and reliable method of contraception.
* Patients with symptoms of significant mental or somatic disease. Inability to cooperate or communicate with the investigator.
* Patients under supervision or guardianship or any patient subject to legal protection

Randomization criteria:

Eligibility criteria (no later than 4 months post-transplantation:

* Renal graft biopsy performed at M3 and adequate histological material sent within the deadline for the determination of EMT.
* Woman of child-bearing potential, even in case of a history of infertility, must use a recognized and reliable method of contraception throughout the study and for 2 months after discontinuing the study treatment.

Non-eligibility criteria (no later than 4 months post-transplantation):

* Acute rejection histologically proven between transplantation and randomization (local reading).
* Acute subclinical rejection diagnosed on the M3 biopsy (except borderline lesions) (local reading).
* Positive anti-donor antibodies at M3.
* Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2 (MDRDa).
* Proteinuria ≥ 1 g/24h.
* Severe hyperlipidemia: total cholesterol ≥ 9.1 mmol/L (≥ 350 mg/dL) and/or triglycerides ≥ 8.5 mmol/L (≥ 750 mg/dL) despite appropriate lipid-lowering therapy.
* Thrombocytopenia (≤ 75000/mm3), absolute neutrophil count (≤ 1500/mm3), leukocytopenia (≤ 2500/mm3) and/or hemoglobin < 8 g/dL.
* ASAT, ALAT or total bilirubin ≥ 3 UNL.
* Medical or surgical condition which in the investigator's opinion might exclude the patient.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- France (21):
  - Novartis Investigative Site, Caen, Cedex
  - Novartis Investigative Site, Angers, France
  - Novartis Investigative Site, Suresnes, France
  - Novartis Investigative Site, Amiens Cedex1
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Vandoeuvre Les Nancys

REFERENCES:
- [Derived] Loupy A, Aubert O, Orandi BJ, Naesens M, Bouatou Y, Raynaud M, Divard G, Jackson AM, Viglietti D, Giral M, Kamar N, Thaunat O, Morelon E, Delahousse M, Kuypers D, Hertig A, Rondeau E, Bailly E, Eskandary F, Bohmig G, Gupta G, Glotz D, Legendre C, Montgomery RA, Stegall MD, Empana JP, Jouven X, Segev DL, Lefaucheur C. Prediction system for risk of allograft loss in patients receiving kidney transplants: international derivation and validation study. BMJ. 2019 Sep 17;366:l4923. doi: 10.1136/bmj.l4923. PMID 31530561

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: EMT+: ≥ 10% tubular cells showing de novo expression of vimentin (or translocation of β catenin if inconclusive) into the cytoplasm EMT-: < 10% tubular cells showing de novo expression of vimentin (or translocation of β catenin if inconclusive) into the cytoplasm
Period: Overall Study
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Started | 36 | 60 | 39 | 59
Exposed | 36 | 60 | 39 | 59
Month 3 (M3) Biopsies | 36 | 59 (1 patient was excluded due to an IF/TA Grade of III at the M3 Biopsy) | 39 | 59
Month 12 (M12) Biopsies | 26 (Only 26 out of 36 participants in this group had graft biopsy that was eligible for analysis.) | 43 | 32 (Only 32 out of 39 participants in this group had graft biopsy that was eligible for analysis.) | 53 (Only 53 out of 59 participants in this group had graft biopsy that was eligible for analysis.)
M3 and M12 Biopsies | 26 (Only 26 out of 36 participants in this group had graft biopsy that was eligible for analysis.) | 43 | 32 (Only 32 out of 39 participants in this group had graft biopsy that was eligible for analysis.) | 53 (Only 53 out of 59 participants in this group had graft biopsy that was eligible for analysis.)
Completed | 27 | 43 | 34 | 54
Not Completed | 9 | 17 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT- | Total
Number analyzed (Participants) | 36 | 60 | 39 | 59 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (10.7) | 46.4 (12.9) | 50.0 (10.0) | 50.7 (11.7) | 49.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 16 | 16 | 66
  Male | 19 | 43 | 23 | 43 | 128
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.3 (4.6) | 26.0 (4.6) | 25.6 (4.0) | 25.3 (4.2) | 25.4 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression of Renal Graft Fibrosis (Primary Comparison - ITT Population
Description: Progression of Interstitial Fibrosis/Tabular Atrophy (IF/TA) is the percentage (%) of participants with an increase >= 1 in IF/TA grade according to Banff (2005 - 2007)according to Epithelial-mesenchymal transition (EMT) profile and by treatment groups.
  Grade I (the better): mild interstitial fibrosis and tubular atrophy (<25% of cortical area) Grade II : moderate interstitial fibrosis and tubular atrophy (26-50% of cortical area) Grade III (the worse) : severe interstitial fibrosis and tubular atrophy (>50% of cortical area)
Time Frame: Month 3 (M3) and Month 12 (M12) post transplantation
Population: ITT population: All patients randomized in the study who received at least one dose of the study treatment. Among the 194 participants in the ITT group, 58 patients in the EMT+ group completed the study providing a graft biopsy for analysis at M3 and M12. The primary comparison concerned only the Certican and the Neoral EMT+ groups.
Measure: Number; unit: Participants
Arm/Group | Certican EMT+ | Neoral EMT+
Number analyzed (Participants) | 26 | 32
Participants
  Participants with an IF/TA grade <= II at M3 | 26 | 31
  Participants with Fibrosis progression, M3 to M12 | 12 | 16

2. Secondary Outcome: Interstitial Fibrosis/Tabular Atrophy (IF/TA)
Description: Incidence and severity of IF/TA according to 2005/2007 Banff classification system grades (grades l to lll). IF/TA grade was assessed during centralized reading according to the Banff 2005/2007 classification comprising grade I (<25%), grade II (25-50%) and grade III (>50% of lesions).
Time Frame: M3 and M12 post transplantation
Population: ITT population: All patients randomized in the study who received at least one dose of the study treatment. Among the 194 participants in the ITT group, 58 patients in the EMT+ group completed the study providing a graft biopsy for analysis at M3 and M12.
Measure: Number; unit: Number of participants
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Number analyzed (Participants) | 26 | 43 | 32 | 53
Number of participants
  Interstitial Fibrosis/Tubular Atrophy (IF/TA) | 13 | 38 | 13 | 44
  IF/TA grade at M3 at grade 1 | 11 | 5 | 17 | 9
  IFTA grade at M3 at grade II | 2 | 0 | 1 | 0
  IF/TA grade at M3 at grade III | 0 | 0 | 1 | 0
  IF/TA grade at M12 at grade 0 | 9 | 20 | 7 | 31
  IT/TA grade at M12 at grade I | 8 | 18 | 15 | 15
  IF/TA grade at M12 at grade II | 6 | 5 | 9 | 6
  IF/TA grade at M12 at grade III | 3 | 0 | 1 | 1

3. Secondary Outcome: Change in Interstitial Fibrosis/Tabular Atrophy (IF/TA) Grade
Description: Difference (M12 - M3) in IF/TA grade. IF/TA grade was assessed during centralized reading according to the Banff 2005/2007 classification comprising grade I (<25%), grade II (25-50%) and grade III (>50% of lesions).
Time Frame: M3 and M12 post transplantation
Population: as for outcome 2
Measure: Number; unit: Number of Participants
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Number analyzed (Participants) | 26 | 43 | 32 | 53
Number of Participants
  Difference in IF/TA grade -1 | 5 | 1 | 7 | 2
  Difference in IF/TA grade 0 | 9 | 21 | 9 | 33
  Difference in IF/TA grade 1 | 7 | 18 | 11 | 13
  Difference in IF/TA grade 2 | 3 | 3 | 5 | 5
  Difference in IF/TA grade 3 | 2 | NA — No analysis done for grade lll for the Certican EMT- arm | 0 | NA — No analysis done for grade lll for the Neoral EMT- arm

4. Secondary Outcome: Risk Factors of IF/TA Progression
Description: Composite factors regarding fibrosis progression at 12 months using a logistic regression model; the parameters initially considered concerned the demographic characteristics of both recipient and donor, transplantation characteristics, hypertension, diabetes, study treatments, immunosuppression, EMT, IF/TA, function at M3, the onset of acute rejection, the presence of anti-donor antibodies at M12, infections and BK virus viremia.
  Arteriolar hyaline thickening is thickening of the walls of arterioles by the deposition of homogeneous pink hyaline material.
  BPAR is biopsy proven acute rejection. TEM progression is the increase ≥ 1 of TEM score between Month 3 and Month 12
Time Frame: M12 post transplantation
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- Yes- Fibrosis Progression: Participants who experienced fibrosis progression based on IF/TA (univariate analysis)
- No- No Fibrosis Progression: Participants who did not experience fibrosis progression based on IF/TA (univariate analysis)
Arm/Group | Yes- Fibrosis Progression | No- No Fibrosis Progression
Number analyzed (Participants) | 67 | 86
Participants
  Donor Sex - Male | 45 | 48
  Donor Sex - Female | 22 | 38
  Donor Age - <=50 years | 28 | 48
  Donor Age - >50 years | 39 | 38
  Expanded Criteria donor: NO | 40 | 63
  Expanded Criteria Donor: Yes | 27 | 23
  Delayed graft function: No | 52 | 76
  Delayed graft function: Yes | 15 | 10
  CC at M3 <50 mL/min/1.73m^2 | 40 | 35
  CC at M3 >=50 mL/min/1.73m^2 (n=67, 85) | 27 | 50
  Mesangial matrix increase at M3 - 0 (n=64, 85) | 59 | 84
  Mesangial matrix (mm) increase at M3: 1 (n=64, 85) | 2 | 1
  Mesangial matrix increase at M3: 2 (n=64, 85) | 3 | 0
  Interstitial fibrosis (ci) at M3: 0 (n=66, 85) | 52 | 55
  Interstitial fibrosis (ci) at M3: 1 (n=66, 85) | 14 | 27
  Interstitial fibrosis (ci) at M3: 2 (n=66, 85) | 0 | 3
  Arteriolar hyaline thickening (ah) at M3: 0 | 36 | 56
  Arteriolar hyaline thickening (ah) at M3: 1 | 15 | 21
  Arteriolar hyaline thickening (ah) at M3: 2 | 10 | 8
  Arteriolar hyaline thickening (ah) at M3: 3 | 6 | 1
  BPAR - No | 55 | 79
  BPAR - Yes | 12 | 7
  TEM Progression fron M3-M12: No (n=67, 83) | 26 | 57
  TEM Progression fron M3-M12: Yes (n=67, 83) | 41 | 26
  TEM Progression fron M3-M12: Missing (n=67, 83) | 0 | 3

5. Secondary Outcome: Change in Percentage of Interstitial Fibrosis (IF) by Numerical Quantification
Description: Percentage of IF measured by numerical quantification. The IF percentage was transposed in grade according to the following rule: grade 0 for an IF % ≤5%, grade I for an IF % ranging from >5% to < 25%, grade II for an IF % ranging from 25 to 50%, grade III for an IF % >50%. Interstitial graft fibrosis has been identified as the primary cause of graft loss following death with a functional graft [3-5].
Time Frame: M3 and M12 post transplantation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of IF
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Number analyzed (Participants) | 26 | 43 | 32 | 53
Percentage of IF
  Percentage of IF at M3 (n=26,43,32,53) | 22.8 (8.9) | 15.9 (7.5) | 23.4 (9.5) | 17.8 (8.2)
  Percentage of IF at M12 (n=24,42,32,53) | 27.6 (12.2) | 20.9 (10.1) | 27.4 (11.5) | 20.4 (9.1)
  Change in Percentage of IF (n=24,42,32,53) | 5.1 (12.4) | 4.9 (12.2) | 3.9 (12.3) | 2.7 (9.7)

6. Secondary Outcome: Number of Participants With Progression of Renal Fibrosis Using Numerical Quantification
Description: Comparisons according to epithelial-mesenchymal transition (EMT) profile and immunosuppressive treatment
Time Frame: M3 to M12 post transplantation
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Number analyzed (Participants) | 26 | 43 | 32 | 53
Participants
  Fibrosis Progression - No (n=24, 42, 31, 53) | 18 | 30 | 19 | 42
  Fibrosis progression - Yes (n=24, 42,31,43) | 6 | 12 | 12 | 11
  Fibrosis progression - Missing (n=24, 42, 31, 53) | 2 | 1 | 0 | 0

7. Secondary Outcome: Number of Participants With Epithelial-mesenchymal Transition (EMT) Status
Description: Incidence and severity of EMT status. EMT status was determined centrally using the graft biopsy taken at 3 months. The result was quickly obtained (within 7 to 15 days) and sent to the company in charge of randomization in order to allocate each patient to a treatment group and to provide the investigator with this information without confirming EMT status.
Time Frame: M3 and M12 post transplantation
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Number analyzed (Participants) | 26 | 43 | 32 | 53
Participants
  EMT Status at M3-Negative (n=26,43,32,53) | 0 | 43 | 0 | 53
  EMT Status at M3- Positive (n=26,43,32,53) | 26 | 0 | 32 | 0
  EMT Status at M3 - Not done (n=26,43,32,53) | 0 | 0 | 0 | 0
  EMT Status at M12- Negative (n=25,41,32,53) | 8 | 24 | 9 | 36
  EMT Status at M12- Positive (n=25,41,32,53) | 17 | 17 | 23 | 17
  EMT Status at M12- Not done (n=25,41,32,53) | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Epithelial-mesenchymal Transition (EMT) Score
Description: Incidence and severity of EMT score. The intensity of EMT markers expression present and detectable in the renal graft at an early stage following transplantation is known as EMT score.
  EMT score 0 (the best): <1 EMT score 1 (the better): 1-10% of tubular atrophy EMT score 2: 10-25% of tubular atrophy EMT score 3: 25-50% of tubular atrophy EMT score 4 (the worst): >50% of tubular atrophy
Time Frame: M3 and M12 post transplantation
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Number analyzed (Participants) | 26 | 43 | 32 | 53
participants
  EMT Score 0 at M3 (n= 26,43,32, 53) | 0 (0.49) | 26 (0.49) | 0 (0.72) | 28 (0.5)
  EMT Score 1 at M3 (n= 26,43,32, 53) | 0 | 17 | 0 | 25
  EMT Score 2 at M3 (n= 26,43,32, 53) | 17 | 0 | 20 | 0
  EMT Score 3 at M3 (n= 26,43,32, 53) | 9 | 0 | 8 | 0
  EMT Score 4 at M3 (n= 26,43,32, 53) | 0 | 0 | 4 | 0
  EMT Score 0 at M12 (n= 25,41,32, 53) | 1 (1.06) | 13 (1.17) | 0 (1.02) | 19 (1.03)
  EMT Score 1 at M12 (n= 25,41,32, 53) | 7 | 11 | 9 | 17
  EMT Score 2 at M12 (n= 25,41,32, 53) | 10 | 11 | 10 | 12
  EMT Score 3 at M12 (n= 25,41,32, 53) | 4 | 4 | 9 | 4
  EMT Score 4 at M12 (n= 25,41,32, 53) | 3 | 2 | 4 | 1
  EMT Missing Score at M12 (n= 25,41,32, 53) | 1 | 2 | 0 | 0

9. Secondary Outcome: Change in EMT Score
Description: Change (M12 - M3) in EMT Score. Progression in EMT score is defined as an increase by >=1 of EMT score from M3 to M12.
  EMT score 0 (the best): <1 EMT score 1 (the better) : 1-10% of tubular atrophy EMT score 2 : 10-25% of tubular atrophy EMT score 3 : 25-50% of tubular atrophy EMT score 4 (the worst): >50% of tubular atrophy
Time Frame: M3 and M12 post transplantation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Number analyzed (Participants) | 26 | 43 | 32 | 53
scores on a scale | -0.3 (1.22) | 0.9 (1.09) | -0.3 (1.05) | 0.6 (0.99)

10. Secondary Outcome: Incidence (Number) of Subclinical Rejections and Borderline Lesions
Description: Incidence of subclinical rejections and borderline lesions with regards to histological evidence of rejection with clinical findings.
  Subclinical rejections: rejection without clinical symptoms which is diagnosed by chance when a graft biopsy is performed.
  Clinically suspected BPAR: rejection suspected because of the presence of clinical symptoms (fever, pain, increase of creatinine) and then confirmed by the graft biopsy.
  Borderline lesions: suspicious for acute T-cell mediated rejection. This category is used when no intimal arteritis is present, but there are foci of tubulitis with minor interstitial infiltration or interstitial infiltration with mild tubulitis.
Time Frame: M3
Population: ITT population: All patients randomized in the study who received at least one dose of the study treatment.
Measure: Number; unit: Participants
Groups:
- Certican: Patients randomized to the Certican® treatment group started this treatment after randomization (which took place 3 to 4 months post-transplantation), preferably in the evening, otherwise the following morning. Patients in the Neoral® treatment group did not receive Certican®.
- Neoral: Between transplantation adn randomization, all patients have received Neoral. Treatment had to be initiated within 24 hours post-transplantation in combination with Myfortic.
Arm/Group | Certican | Neoral
Number analyzed (Participants) | 69 | 85
Participants
  Subclinical rejections-No (n=68, 84) | 67 | 84
  Subclinical rejections- Yes (n=68, 84) | 1 | 0
  Subclinical rejections- missing (n=68, 84) | 1 | 1
  Clinically suspected BPAR - No (N=68, 84) | 68 | 84
  Clinically suspected BPAR - Yes (N=68, 84) | 0 | 0
  Clinically suspected BPAR - Missing (N=68, 84) | 1 | 1
  Borderline lesions - No (n=68,84) | 62 | 71
  Borderline lesions - Yes (n=68,84) | 6 | 13
  Borderline lesions - Missing (n=68,84) | 1 | 1

11. Secondary Outcome: Change From Baseline (M3) in Estimated Glomerular Filtration Rate (eGFR)
Description: eGFR was calculated according to the abbreviated Modification of Diet in Renal Disease (MDRD) Formula and creatinine clearance according to the Cockcroft-Gault formula (mL/min/1.73m²).
  LOCF = Last observation carried forward
Time Frame: M3 (baseline) to M12 post transplantation
Population: ITT population: All patients randomized in the study who received at least one dose of the study treatment.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2
Groups:
- Neoral: Between transplantation and randomization, all patients have received Neoral®. Treatment had to be initiated within 24 hours post-transplantation in combination with Myfortic®.
Arm/Group | Certican | Neoral
Number analyzed (Participants) | 71 | 87
mL/min/1.73m^2
  without imputation | 6.99 (1.66) | 2.54 (1.5)
  imputation by LOCF(96, 97) | 5.96 (1.39) | 2.15 (1.37)

12. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR) at M12 From Baseline (M3) - ANCOVA Model
Description: The average patient renal function was evaluated on the basis of eGFR was calculated according to the abbreviated MDRD formula and creatinine clearance according to the Cockcroft-Gault formula (mL/min/1.73m²).
Time Frame: Baseline (M3), M12
Population: ITT population: All patients randomized in the study who received at least one dose of the study treatment.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m²
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Number analyzed (Participants) | 27 | 44 | 34 | 53
mL/min/1.73m²
  without imputation | 8.6 (15.21) | 5.6 (18.73) | 1.5 (9.49) | 3.8 (10.99)
  imputation by LOCF (36, 60, 39, 58) | -11.9 (27.78) | 27.3 (138.44) | 5.1 (40.80) | -4.9 (29.09)

13. Secondary Outcome: Change in Urine Protein/Creatinine Ratio (Without Imputation)
Description: One of the factors associated with EMT progression between M3 and M12 according to univariate analysis (ITT biopsies M3 & M12).
Time Frame: Month 3 (baseline), Month 12
Population: ITT population: All patients randomized in the study who received at least one dose of the study treatment.
Measure: Mean (Standard Deviation); unit: mg/mmol
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Number analyzed (Participants) | 17 | 28 | 19 | 36
mg/mmol | 44.4 (188.99) | 3.5 (48.37) | 16.0 (41.53) | 29.8 (189.41)

14. Secondary Outcome: Treatment Failures
Description: A treatment failure is defined as biopsy proven acute rejection (BPAR), a graft loss, a death or a loss to follow up. It was assessed between randomization and 6 and 12 months post-transplantation.
Time Frame: M6 and M12 post transplantation
Population: ITT population: All patients randomized in the study who received at least one dose of the study treatment.
Measure: Number; unit: Number of Participants
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Number analyzed (Participants) | 36 | 60 | 39 | 59
Number of Participants
  M6: Treatment Failure- No | 33 | 52 | 39 | 59
  M6: Treatment Failure- Yes | 3 | 8 | 0 | 0
  M12: Treatment Failure- No | 29 | 42 | 36 | 56
  M12: Treatment Failure- Yes | 7 | 18 | 3 | 3
  M6: BPAR - No | 33 | 52 | 39 | 59
  M6: BPAR -Yes | 3 | 8 | 0 | 0
  M12: BPAR - No | 29 | 43 | 37 | 56
  M12: BPAR - Yes | 7 | 17 | 2 | 3
  M6: Graft Loss - No | 36 | 60 | 39 | 59
  M6: Graft Loss - Yes | 0 | 0 | 0 | 0
  M12: Graft Loss - No | 35 | 56 | 38 | 59
  M12: Graft Loss - Yes | 1 | 4 | 1 | 0
  M6: Death - No | 36 | 60 | 39 | 59
  M6: Death - Yes | 0 | 0 | 0 | 0
  M12: Death - No | 36 | 60 | 39 | 59
  M12: Death - Yes | 0 | 0 | 0 | 0
  M6: Loss to follow-up - No | 36 | 60 | 39 | 59
  M6: Loss to follow-up - Yes | 0 | 0 | 0 | 0
  M12: Loss to follow-up - No | 36 | 59 | 39 | 59
  M12: Loss to follow-up - Yes | 0 | 1 | 0 | 0

15. Secondary Outcome: Type of Biopsy Proven Acute Rejection (BPAR)
Description: A biopsy proven acute rejection (BPAR) is defined as a biopsy graded IA, IB, IIA, IIB or III as per 2005/2007 Banff histological classification system.
  Biopsy graded IA: Significant interstitial infiltration (> 25% of parenchyma) and foci of moderate tubulitis (> 4 mononuclear cells/tubular cross section or group of 10 tubular cells).
  Biopsy grade IB: Significant interstitial infiltration (> 25% of parenchyma) and foci of severe tubulitis (> 10 mononuclear cells/tubular cross section or group of 10 tubular cells).
  Biopsy grade IIA: Mild to moderate intimal arteritis. Biopsy graded IIB: Severe intimal arteritis comprising > 25% of the lumenal area.
  Biopsy graded III: Transmural (full vessel wall thickness) arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells (with accompanying lymphocytic inflammation).
Time Frame: M6 and M12 post transplantation
Population: ITT population: All patients randomized in the study who received at least one dose of the study treatment.
Measure: Number; unit: Participants
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Number analyzed (Participants) | 36 | 60 | 39 | 59
Participants
  Cellular AR - No | 30 | 46 | 38 | 58
  Cellular AR - Yes | 6 | 14 | 1 | 1

16. Secondary Outcome: Severity of BPAR
Description: as for outcome 15
Time Frame: M6 and M12 post transplantation
Population: ITT population: All patients randomized in the study who received at least one dose of the study treatment.
Measure: Number; unit: Participants
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Number analyzed (Participants) | 36 | 60 | 39 | 59
Participants
  M6: Banff type Grade IA | 0 | 2 | 0 | 0
  M6: Banff type Grade IB | 0 | 4 | 0 | 0
  M6: Banff type Grade IIA | 1 | 0 | 0 | 0
  M6: Banff type Grade IIB | 0 | 1 | 0 | 0
  M6: Banff type Grade III | 0 | 0 | 0 | 0
  M12: Banff type Grade IA | 2 | 7 | 1 | 0
  M12: Banff type Grade IB | 2 | 5 | 0 | 0
  M12: Banff type Grade IIA | 1 | 1 | 0 | 1
  M12: Banff type Grade IIB | 0 | 1 | 0 | 0
  M12: Banff type Grade III | 0 | 0 | 0 | 0

17. Secondary Outcome: Incidence (Number) of BPAR
Description: A biopsy proven acute rejection (BPAR) is defined as a biopsy graded IA, IB, IIA, IIB or III as per 2005/2007 Banff histological classification system.
Time Frame: M6 and M12 post transplantation
Population: ITT population: All patients randomized in the study who received at least one dose of the study treatment.
Measure: Number; unit: Number of participants
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Number analyzed (Participants) | 36 | 60 | 39 | 59
Number of participants
  M6 - No | 33 | 52 | 39 | 59
  M6 - Yes | 3 | 8 | 0 | 0
  M12 - No | 29 | 43 | 37 | 56
  M12 - Yes | 7 | 17 | 2 | 3

18. Secondary Outcome: Incidence (Number) of Participants With Graft Losses
Description: If a participant underwent a graft nephrectomy, then the day of nephrectomy was considered as the day of graft loss.
Time Frame: M6 and M12 post transplantation
Population: ITT population: All patients randomized in the study who received at least one dose of the study treatment.
Measure: Number; unit: Participants
Arm/Group | Certican EMT+ | Certican EMT- | Neoral EMT+ | Neoral EMT-
Number analyzed (Participants) | 36 | 60 | 39 | 59
Participants
  M6 - No | 36 | 60 | 39 | 59
  M6 - Yes | 0 | 0 | 0 | 0
  M12 - No | 35 | 56 | 38 | 59
  M12 - Yes | 1 | 4 | 1 | 0

ADVERSE EVENTS:
Arm/Group | Neoral | Certican
Serious Adverse Events (participants affected / at risk) | 39/98 | 46/96
Other Adverse Events (participants affected / at risk) | 59/98 | 59/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoral (N=98) | Certican (N=96)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 0 | 2
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Dental necrosis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Gastritis (Gastrointestinal disorders) | 1 | 0
Hernial eventration (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 1
Chills (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 5
Sudden death (General disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Amyloidosis (Immune system disorders) | 1 | 0
Kidney transplant rejection (Immune system disorders) | 0 | 4
Transplant rejection (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Bacillus infection (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 3 | 2
Bronchitis (Infections and infestations) | 0 | 2
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 2
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Eye infection toxoplasmal (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis yersinia (Infections and infestations) | 0 | 1
Hepatic cyst infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Polyomavirus-associated nephropathy (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 3
Pyelonephritis acute (Infections and infestations) | 1 | 3
Renal cyst infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Transplant abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 4
Viral pharyngitis (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 | 0
Graft loss (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 2
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 2
Blood pressure increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Neurosis (Psychiatric disorders) | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 4 | 2
Renal tubular disorder (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Capillaritis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Iliac artery stenosis (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neoral (N=98) | Certican (N=96)
Anaemia (Blood and lymphatic system disorders) | 6 | 7
Leukopenia (Blood and lymphatic system disorders) | 7 | 2
Neutropenia (Blood and lymphatic system disorders) | 6 | 6
Aphthous stomatitis (Gastrointestinal disorders) | 3 | 17
Diarrhoea (Gastrointestinal disorders) | 3 | 7
Gingival hypertrophy (Gastrointestinal disorders) | 8 | 0
Oedema peripheral (General disorders) | 17 | 14
Bronchitis (Infections and infestations) | 6 | 5
Cytomegalovirus infection (Infections and infestations) | 7 | 2
Urinary tract infection (Infections and infestations) | 5 | 7
Dyslipidaemia (Metabolism and nutrition disorders) | 6 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 7
Hypertension (Vascular disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.